CLINICAL TRIAL: NCT07084207
Title: REGEN: A Prospective, Randomized, Open Label Study to Expand the Use of Symani® Surgical System for Peripheral Nerve Repair
Brief Title: A Study to Expand the Use of Symani® Surgical System for Peripheral Nerve Repair
Acronym: REGEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MMI (Medical Microinstruments, Inc.) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDC-00146
Record Dates: First submitted 2025-07-03; First posted 2025-07-24 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Nerve Injury; Peripheral Nerve Injuries
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Robotic-Assisted Surgery (RAS) group (Active Comparator)
  Interventions: Device: Symani® Surgical System
- Manual Surgery (MS) group (Active Comparator)
  Interventions: Procedure: Manual Surgery

INTERVENTIONS:
Device: Symani® Surgical System — Robotic-assisted surgery consists of participants who undergo nerve coaptation with the Symani Surgical System, according to the Instruction for Use (IFU). In order for the surgery to be considered a robotic assisted surgery, the participants must be randomized to the RAS group which will include:
  * Participants where all nerve coaptations were performed entirely with Symani.
  * Participants who underwent a hybrid procedure, where a coaptation was commenced using Symani but a switch to manual suturing occurred during the procedure
  Other Names: RAS
  Arms: Robotic-Assisted Surgery (RAS) group
Procedure: Manual Surgery — Manual surgery consists of participants who undergo nerve coaptation through manual techniques by a surgeon using handheld instruments without robotic assistance. In order for the surgery to be considered a manual surgery, the participants must be randomized to the MS group which will include:
  * Participants where all nerve coaptations were performed entirely manually.
  * Participants who underwent a hybrid procedure, where a coaptation was commenced using manual suturing but a switch to Symani occurred during the procedure.
  Other Names: MS
  Arms: Manual Surgery (MS) group

SUMMARY:
The objective of this study is to evaluate the Symani System's safety and effectiveness for microsurgical nerve coaptation, following nerve injuries to the hand.

This study will include participants with traumatic sensory nerve lesions of a finger nerve distal to the carpal tunnel who are treated with nerve suturing.

The primary effectiveness endpoint is the two-point discrimination (2PD) test, at 6-months post index procedure.

The primary safety endpoint is the intraoperative serious adverse event rate.

ELIGIBILITY:
Pre-Operative

Inclusion Criteria:

1. Adults, at the time of nerve injury aged from 18 to 70 years
2. Patient agrees to participate in the study, returns for all required follow-up visits, and has willingly provided written informed consent after receiving all information related to the study and its requirements
3. Complete loss of a nerve-specific receptive field of the finger
4. Patient with a clinical indication for a microsurgical nerve coaptation in nerve injury that can be repaired by end-to-end suturing
5. Patient with traumatic transection of one or more digit nerves distal to the carpal tunnel with sensory autonomous innervation areas on the finger or thumb tips
6. Investigator considers candidate acceptable for either conventional epineural suturing or robotic-assisted epineural suturing
7. The injury was treated within 10 days

Exclusion Criteria:

1. Patients who are not capable and/or unwilling to provide informed consent
2. Clinically significant cardiovascular, digestive, respiratory, endocrine, liver or central nervous system disorders, previous mental disorders, or other disorders that may significantly affect the data collection or the ability to comply with the protocol per the investigators' discretion.
3. Currently enrolled in any other investigational clinical studies that the investigator believes may impact patient safety or outcomes
4. Patients belonging to vulnerable populations, such as pregnant women, or patients ineligible to participate for other reasons in the judgement of the investigator
5. Indication for bilateral nerve repair
6. Known impaired sensibility of the injured finger
7. Patients with implanted pacemaker
8. Replantation which includes bones

Intra-Operative Inclusion Criteria

Individuals will be included in the study if the following criteria are met intraoperatively:

1. Verification of a sensory nerve lesion without a gap and presence of a nerve that could be sutured in end-to-end fashion Intra-Operative Exclusion Criteria

Individuals will be excluded from participating in this study if any of the following criteria are met intraoperatively:

1. Any presenting condition discovered intraoperatively that, in the opinion of the investigator, would

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2026-12-18 (Estimated); Study Completion 2027-12-18 (Estimated)

PRIMARY OUTCOMES:
Two-point discrimination (2PD) test, at 6-months post index procedure. | From participants index procedure through 6-months post index procedure
  The primary effectiveness endpoint is the two-point discrimination (2PD) test, at 6-months post index procedure.
  The two-point discrimination test is a sensory test used to assess the ability of the patient to distinguish between two distant points of touch on the skin. The test measures the minimum distance between two stimulus points on the skin, which are perceived as distinct points. This endpoint will be evaluated at 6-months post index procedure.
Intraoperative serious adverse event rate | The duration of the participants index procedure.
  The primary safety endpoint is the intraoperative serious adverse event rate.
  The incidence of SAEs occurring during the intra-operative period will be presented. In addition, each participant will be categorized as 'had any SAEs in the intra-operative period' Yes or No. The proportion of participants who experienced any SAEs in the intra-operative period will be presented with exact confidence limits. The difference between groups will also be presented with exact confidence limits.

SECONDARY OUTCOMES:
Two-point discrimination test at 3 and 12-months post index procedure | From participants index procedure through 3-months and 12-months post-index procedure
  The two-point discrimination test (2PD) will be assessed at 3, 6, 12-months post-surgery. It will be measured in mm.
  Descriptive statistics will be presented by surgical group and timepoint. A mixed model for repeated measures (MMRM) will be fitted with 2PD (mm) as the outcome and surgical group, timepoint and surgical group*timepoint as fixed effects. Timepoint will be included as a repeated term (subject=participant) to acknowledge the repeated measures in the study (i.e. a participant will have data for 3, 6, and 12-months). Nerve will also be included as a repeated term (subject=participant) to acknowledge that a participant may have more than one nerve involved. Other terms may be included, as defined in the SAP.
  From the model the least squares means (LSM) for each surgical group at each timepoint will be presented with confidence limits (CLs). In addition, the difference in LSMs between groups at each timepoint will be presented with CL.
Ten Test on sensitivity at 3, 6 and-12 months post index procedure | From participants index procedure through 3-months and 12-months post-index procedure
  Ten Test is defined as the assessment of sensory function in the injured and contralateral nerves, using a scale from 0 (no sensitivity) to 10 (full sensitivity). The results will be compared between the injured and contralateral nerves to evaluate sensory function. This endpoint will be evaluated at 3-months, 6-months and 12-months post-index procedure.
Sensory reinnervation assessment (Semmes-Weinstein monofilament method) at 3, 6 and-12 months post index procedure | From participants index procedure through 3-months, 6-months and 12-months post-index procedure
  Sensory Reinnervation is defined as the smallest filament detected on both the affected and contralateral nerves using the Semmes-Weinstein Monofilament Test. The endpoint will be evaluated at 3-months, 6-months, and 12-months post-index procedure
Gross hand strength assessment (Jamar Dynamometer) at 3, 6 and 12-months after post procedure | From participants index procedure through 3-months, 6-months and 12-months post-index procedure
  Gross Hand Strength is defined as the measurement of hand strength using a dynamometer, recorded in kilograms (kg). Strength will be assessed for both the injured hand and the contralateral hand, with results recorded for each hand. This endpoint will be evaluated at 3-months, 6-months and 12-months post-index procedure.
Thumb strength assessment (Jamar Dynamometer) at 3, 6 and 12-months post index procedure | From participants index procedure through 3-months, 6-months and 12-months post-index procedure
  Thumb Strength Assessment is defined as the measurement of thumb strength using a Jamar Dynamometer, recorded in kilograms (kg). Strength will be assessed for both the injured hand and the contralateral hand. This endpoint will be evaluated at 3-months, 6-months and 12-months post-index procedure.
Range of motion of the injured finger in flexion and extension in comparison with the unaffected side at 3, 6 and 12-months post index procedure | From participants index procedure through 3-months, 6-months and 12-months post-index procedure
  Range of Motion (ROM) is defined as whether the injured finger achieves full flexion and extension compared to the unaffected side. This endpoint will be evaluated at 3-months, 6-months, and 12-months post-index procedure.
Kapandji Score at 3, 6 and 12-months after post procedure | From participants index procedure through 3-months, 6-months and 12-months post-index procedure
  The Kapandji Score will be defined as a measure of thumb opposition, with scores ranging from 0 to 10, where a higher score indicates better thumb mobility and function. Results from each time point will be used to assess changes in thumb opposition and overall hand function. Assessments will be made at 3-months, 6-months and 12-months post-index procedure
DASH questionnaire at 3, 6 and 12-months post index procedure | From participants index procedure through 3-months, 6-months and 12-months post-index procedure
  The Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire will be used to assess the participants' upper limb function, specifically related to the arm, shoulder, and hand. It measures the severity of symptoms and the impact of musculoskeletal disorders or injuries on daily activities. The DASH questionnaire consists of 30 items covering aspects like physical function, symptoms, and social or work-related limitations. The score ranges from 0 to 100. A higher score indicating greater disability or dysfunction. This questionnaire will be administered to each participant either on paper or electronically at the 3-month, 6-month, and 12-month follow-up visits. The DASH questionnaire will be completed individually by each participant.
  The DASH Questionnaire will assess the physical function and symptoms (such as pain and weakness) of the arm, shoulder, and hand, evaluating the participant's ability to perform daily activities. These functio

CONTACTS AND LOCATIONS:
Locations (1):
- BG Klinik Ludwigshafen, Ludwigshafen, Germany